CLINICAL TRIAL: NCT05023148
Title: Comparison Therapeutic Effects Between Electroacupuncture and Thread Embedded Acupuncture in Obese Patients With Dietary Intervention
Brief Title: Comparison of Electroacupuncture and Thread Embedded Acupuncture With Dietary Intervention in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Cindy Notonegoro, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-05-0530
Record Dates: First submitted 2021-08-22; First posted 2021-08-26 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Obesity
Keywords: electroacupuncture; thread embedded acupuncture; obese; dietary intervention
MeSH Terms: conditions — Obesity | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: There are two groups of intervention. The first group is getting electroacupuncture treatment and the second group is getting thread embedded acupuncture treatment.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and laboratory analyst do not know which group that participants was assigned in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture with dietary intervention (Active Comparator): Acupoints stimulation with an electric stimulator on CV12 Zhongwan, CV9 Shuifen, CV6 Qihai, CV4 Guanyuan, ST25 Tianshu bilateral, SP15 Daheng bilateral, ST40 Fenglong bilateral using continuous 2 Hz for 30 minutes. Therapy sessions are three times a week for four weeks (total 12 times).
  Dietary intervention means reducing 500 calories from usual calorie consumptions and will be done twice, at the beginning and 2 weeks after.
  Interventions: Procedure: Electroacupuncture
- Thread embedded acupuncture with dietary intervention (Active Comparator): Acupoints stimulation by embedding PDO thread in CV12 Zhongwan penetrating to CV9 Shuifen using 27G x 60 mm, CV4 Guanyuan penetrating to CV6 Qihai using 27G x 40 mm, ST25 Tianshu penetrating to SP15 Daheng using 27G x 40 mm, and perpendicular in ST40 Fenglong bilateral using 31G x 25 mm. Therapy will be done only once.
  Dietary intervention means reducing 500 calories from usual calorie consumptions and will be done twice, at the beginning and 2 weeks after.
  Interventions: Procedure: Thread embedded acupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Stimulating acupoints using electric stimulator
  Arms: Electroacupuncture with dietary intervention
Procedure: Thread embedded acupuncture — Stimulating acupoints using thread embedded
  Arms: Thread embedded acupuncture with dietary intervention

SUMMARY:
The purpose of this study is to compare the effectiveness between electroacupuncture treatment with dietary intervention and thread embedded acupuncture with dietary intervention in reducing body weight, waist circumference, and leptin level in obese patients.

DETAILED DESCRIPTION:
The purpose of this study is to describe reducement in body weight, waist circumference, and leptin level in obese patients with dietary intervention and electroacupuncture or dietary intervention with thread embedded acupuncture. It is also to analyze mean differences of body weight, waist circumference, and leptin level in obese patients between the two interventions. The results of the study expected to be used as an operating standard procedure for obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60 years
* Obese with Body Mass Index (BMI) 25 - 35 kg/m^2
* Waist circumference male > 90 cm and female > 80 cm
* Willing to participate in the study by signing an informed consent
* Willing to follow the study process until it is finished

Exclusion Criteria:

* Pregnancy
* Post partum < 6 months
* Diabetes (Blood glucose POCT (Point of Care Testing) >= 200 mg/dl)
* Hypertension (Blood pressure >= 140/90 mmHg)
* Fever > 38^C
* Has a history of contraindication for electroacupuncture such as history of heart diseases, pace maker, arrhythmia
* Has a history of contraindication for thread embedded acupuncture such as allergy of PDO (Polydioxanone), blood clotting disorder, consumption of anticoagulant drugs, local infection or wound on embedded site
* Has a history of weight loss drugs consumption (such as orlistat, phentermine, diethylpropion) or slimming supplements (green tea, jati belanda/Guazuma ulmifolia) for the last 25 hours.
* History of liver disease, kidney disease
* Has had acupuncture therapy for obesity in the last six months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Body weight | 1 month
  Participants' body weight in kilograms
Waist circumference | 1 month
  Waist circumference is measured at the end of several consecutive natural breaths, at the level parallel to the floor, midpoint between the top of the iliac crest and the lower margin of the last palpable rib in the midaxillary line
Leptin level | 1 month
  Plasma leptin examination using ELISA method

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Notonegoro, dr., Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No